CLINICAL TRIAL: NCT06000150
Title: Characteristics of Trachomatous Corneal Opacity in Fayoum University Hospital
Acronym: Trachoma
Status: Completed | Type: Observational
Sponsor: Omar Said (Other)
Responsible Party: Sponsor-Investigator, Omar Said, Assistant Professor of Ophthalmology, Fayoum University
Organization: Fayoum University (Other)
Other Study IDs: M356
Record Dates: First submitted 2023-08-12; First posted 2023-08-21 (Actual); Last update posted 2023-08-21 (Actual); Status verified 2023-08

CONDITIONS: Corneal Opacity
MeSH Terms: conditions — Corneal Opacity | interventions — Corneal Topography

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 6 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

INTERVENTIONS:
Diagnostic Test: Corneal topography — AS-OCT,PENTACAM

SUMMARY:
The purpose of this study is to assess the characteristics of trachomatous corneal opacity in patients with signs of trachoma using Anterior segment Optic coherence tomography and Pentacam

DETAILED DESCRIPTION:
After approval of the local institutional ethics committee and local institutional review board, patient presented to Fayoum University Hospital was examined for corneal opacity with signs of trachoma after a detailed informed consent was signed by eligible patients and investigated by Anterior Segment Optic coherence Tomography and Pentacam.

Descriptive statistics were presented in the form of mean and standard deviation for numerical variables while numbers and percentages are used for the categorical variables.

Paired samples t-test was used to study anterior segment Optic Coherence tomography and pentacam in evaluating corneal thickness. Bland-Altman plot was used to study the agreement between the two methods IBM SPSS version 28 for Windows software was used for the analysis and Stata 16 was used for the Bland-Altman plot. A p-value of < 0.05 was considered significant.

ELIGIBILITY:
Inclusion Criteria:

* patients with corneal opacity accompanied by signs of trachoma

Exclusion Criteria:

* corneal opacity due other causes
* history of corneal surgery

Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Patients with trachomatous corneal opacity
Sampling Method: Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2022-02-01 (Actual); Primary Completion 2022-08-30 (Actual); Study Completion 2022-08-30 (Actual)

PRIMARY OUTCOMES:
Corneal imaging | we will recruit patients who meer the inclusion criteria during the study period february-August 2022
  AS-OCT and PENTACAM in patients with trachomatous corneal opacity

CONTACTS AND LOCATIONS:
Locations (1):
- Fayoum University, Al Fayyum, Egypt

IPD SHARING:
Plan to Share IPD: Undecided